CLINICAL TRIAL: NCT04720209
Title: Taking AIM at Breast Cancer: Targeting Adiposity and Inflammation With Movement to Improve Prognosis in Breast Cancer Survivors
Brief Title: Taking AIM at Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-172
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
Keywords: Breast Cancer; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Circuit-style aerobic and resistance Exercise(CARE) (Experimental): This research study involves exercise. Participants in this study will be assigned to one of 2 exercise groups, undergo three (voluntary) biopsies of fat tissue, and participate in 7 testing visits and 48 exercise training visits. Participation is expected to last 12 months.
  -16 weeks of circuit-style aerobic and resistance exercise
  Interventions: Other: CARE
- Traditional Aerobic Resistance Exercise (TARE) (Experimental): This research study involves exercise. Participants in this study will be assigned to one of 2 exercise groups, undergo three (voluntary) biopsies of fat tissue, and participate in 7 testing visits and 48 exercise training visits. Participation is expected to last 12 months
  - 16 weeks of traditional aerobic and resistance exercise
  Interventions: Other: TARE
- Home-Based Stretching (Active Comparator): Attention Control for 16 weeks home-based stretching
  -structured home-based stretching program, participants will be asked to maintain their current activity level for the 4-month study duration, and will be offered the CARE program upon study completion
  Interventions: Other: Home-Based Stretching

INTERVENTIONS:
Other: CARE — CARE is a 16-week, supervised, periodized AE and RE program performed in a circuit fashion 3 days/week on-site
  Arms: Circuit-style aerobic and resistance Exercise(CARE)
Other: TARE — TARE is a 16- week, supervised AE and RE program consisting of three sessions per week on-site
  Arms: Traditional Aerobic Resistance Exercise (TARE)
Other: Home-Based Stretching — This group will perform a home-based program of the same stretches utilized in the CARE and TARE groups.
  Arms: Home-Based Stretching

SUMMARY:
The purpose of this research is to determine whether a 16-week exercise program for individuals with breast cancer and have completed treatment (i.e., surgery, chemotherapy, or radiation) for breast cancer will decrease inflammation in fat tissue.

DETAILED DESCRIPTION:
This study is about using different types of exercise to reduce inflammation in fat tissue in an effort to minimize the risk of cancer recurrence related to being overweight or obese. The investigators hope to learn whether participating in a specific exercise program can cause inflammation in the fat tissue to decrease.

The names of the study interventions involved in this study are:

* Circuit-style aerobic and resistance exercise (CARE)
* Traditional aerobic and resistance exercise (TARE)

The research study procedures include screening for eligibility, and study treatment including evaluations and follow up visits.

The study treatment will be for 4 months and participants will followed for 8 months.

The total time for participation in this study will be about 12 months. It is expected that about 300 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with breast cancer (all stages excluding stage IV), low grade disease positive for estrogen and progesterone receptors
* Over the age of 18 years; children under the age of 18 will be excluded due to rarity of disease
* The effects of exercise on the developing fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately. Patients must undergo a pregnancy test via urine strip that will be covered and provided by the PI. Urine strips will be utilized over bloodwork for cost effectiveness. Urine tests will be distributed once before DEXA scans.
* Are centrally obese with the following criteria[57] (determined by study team at eligibility screening): BMI >30 kg/m2 (calculated using height and weight; an upper limit BMI will not be set; we will rely on obtaining physicians' clearance to assess full eligibility) or body fat >30% (estimated by bioelectrical impedance), and waist circumference >35 in.
* Have undergone a lumpectomy or mastectomy.
* If cancer treatment included neoadjuvant or adjuvant chemotherapy and/or radiation therapy, participant must have received and completed treatment.
* Speak English
* Is in breast cancer remission with no detectable disease present
* Able to initiate a supervised exercise program (free from any cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity)
* Free from history of chronic disease including uncontrolled diabetes, hypertension or thyroid disease.
* Have not experienced a weight reduction ≥10% within the past 6 months
* Currently participate in less than 60 minutes of structured exercise/week
* No planned reconstructive surgery with flap repair during trial and follow-up period
* May use adjuvant endocrine therapy, trastuzumab or pertuzumab if use will be continued for duration of study intervention
* Does not smoke (no smoking during previous 12 months)
* Willing to travel to Dana-Farber Cancer Institute
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection, uncontrolled diabetes, hypertension or thyroid disease
* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* Patients with other active malignancies are ineligible for this study.
* Patients with metastatic disease
* Is not centrally obese as defined above
* Has not completed surgery, chemotherapy, or radiation treatment associated with their diagnosis
* History of any musculoskeletal, cardiorespiratory or neurological diseases that preclude the participation in exercise
* Participates in more than 60 minutes of structured exercise/week
* Is planning reconstructive surgery with flap repair during trial and follow-up period
* Currently smokes
* Is unable to travel to the exercise facilities
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Decrease in adipose tissue levels of inflammation. | 16 Weeks
  Adipose tissue inflammation will be assessed by measuring: M1 and M2 adipose tissue macrophages (ATMs)
Decrease in adipose tissue levels of inflammation. | 16 weeks
  Adipose tissue inflammation will be assessed by measuring: leptin, adiponectin, IL-6 and IL-8
Decrease in adipose tissue levels of inflammation. | 16 weeks
  Adipose tissue inflammation will be assessed by measuring: hs-CRP and TNF-a

SECONDARY OUTCOMES:
4-month CARE intervention on sarcopenic obesity. | 16 Weeks
  sarcopenic obesity will be assessed via dual energy X-ray absorptiometry using a validated equation.

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Dieli-Conwright, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu